CLINICAL TRIAL: NCT03267979
Title: Assessing Pain in the Postoperative Period by Automatically Measuring the Variation Coefficient of Pupillary Diameter: PREVANS Study
Acronym: PREVANS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRBN402014/CHUSTE; CNIL (Other: 1800890)
Record Dates: First submitted 2017-08-25; First posted 2017-08-31 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Anesthesia, General
Keywords: pain assessment; pupillary diameter; variation coefficient of pupillary diameter; pain self assessment; video-pupillometer; electrocardiogram; analgesic treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients have a surgical operation (Other): Patients have a surgical operation and have received analgesic treatment. One hour after the end of surgical patients will have electrocardiogram and video-pupillometer.
  Interventions: Other: Video-pupillometer; Other: Electrocardiogram

INTERVENTIONS:
Other: Video-pupillometer — Video-pupillometer will be performed. In this study data will be collected and analyzed.
  Other Names: Algiscan
Other: Electrocardiogram — Electrocardiogram will be performed. In this study data will be collected and analyzed.

SUMMARY:
Different pain assessment methods have been proposed to evaluate analgesic efficacy after surgical operation. Pain is a subjective phenomenon. Patient did his pain self assessment. But, cooperation of the patient is limited by cultural differences, language barriers or residual effect of products used while general anesthesia.

A lot of study were conducted to demonstrate and to quantify the pain after an operation. The aim will be dose analgesic treatment better without cooperation of the patient.

This sudy concerns patients on the post anesthesia care units one hour after their arrival. They will have electrocardiogram and video-pupillometer.

DETAILED DESCRIPTION:
Primary objective is to compare Variation Coefficient of Pupillary Diameter (VCPD) obtained during a light flash and pain assessment realized thanks to Visual Analog Scale (VAS). Too, Variation Coefficient of Pupillary Diameter (VCPD) with electrocardiogram will be measured to demonstrate a correlation between the three parameters.

ELIGIBILITY:
Inclusion Criteria:

* Major patients
* Patients fluent in French
* Patient admitted on the post anesthesia care units

Exclusion criteria:

* Patients operated for all types of surgery except for heart, intra-cerebral, and ophthalmologic surgeries
* Emergency operation
* Heart rhythm disorders
* Pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2014-11-02 (Actual); Primary Completion 2015-03-31 (Actual); Study Completion 2015-03-31 (Actual)

PRIMARY OUTCOMES:
Correlation between pupillary diameter (PD) and pain assessment | 1 hour post surgery
  Correlation between pupillary diameter (PD) and pain in the post-operative period.
  PD will be measured by video-pupillometer. Pain will be measured by Visual Analog Scale (VAS).

SECONDARY OUTCOMES:
Correlation between pupillary diameter (PD) and heart rate | 1 hour post surgery
  Correlation between pupillary diameter (PD) and heart rate in the post-operative period.
  Heart rate will be measured by electrocardiogram.

CONTACTS AND LOCATIONS:
Overall Officials: David CHARIER, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Charier D, Vogler MC, Zantour D, Pichot V, Martins-Baltar A, Courbon M, Roche F, Vassal F, Molliex S. Assessing pain in the postoperative period: Analgesia Nociception IndexTMversus pupillometry. Br J Anaesth. 2019 Aug;123(2):e322-e327. doi: 10.1016/j.bja.2018.09.031. Epub 2019 Jan 26. PMID 30915996